CLINICAL TRIAL: NCT06067035
Title: Imaging of Small-vessel Liver Tumours
Brief Title: Hepatic Small Vessel Neoplasm
Acronym: IMAHEP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220863
Record Dates: First submitted 2023-09-22; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Hepatic Small Vessel Neoplasm
Keywords: Vascular tumors; Hepatic imaging; Neoplasm
MeSH Terms: conditions — Vascular Neoplasms; Neoplasms | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Imaging — Imaging data from patients with small-vessel liver tumours will be compared with histological data.
  Other Names: surgical specimen

SUMMARY:
Small-vessel hepatic tumor is a new tumor entity of vascular origin, described in 2016 by Gill et al, in a series of 17 patients. This rare lesion is difficult to diagnose on imaging because it shares a common radiological semiology with several other differential diagnoses ranging from benign hepatic angioma to more aggressive lesions such as angiosarcoma.

DETAILED DESCRIPTION:
The aim of our study is to enable the imaging diagnosis of a new entity: small vessel hepatic tumor in order to improve diagnostic management.

ELIGIBILITY:
Inclusion Criteria:

* Histological evidence of a small vessel hepatic tumor either on biopsy or surgical specimen
* Cross-sectional imaging before the biopsy or pre-operatively (CT, MRI)

Exclusion Criteria:

* Patient under guardianship or curators

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with small-vessel liver tumours
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Imaging findings | 12 months
  Aspect on US Ultrasound Scan (US)

SECONDARY OUTCOMES:
Pathological examination | 12 months
  tumors
Biology | 12 months
  bilirubin and alkaline phosphatase rate

CONTACTS AND LOCATIONS:
Overall Officials: MAITE LEWIN, MD, PHD, Study Director — APHP

IPD SHARING:
Plan to Share IPD: No